CLINICAL TRIAL: NCT03827447
Title: Randomized Double Blind Placebo Controlled Trial for the Treatment of NAAT(+)/Toxin EIA(-) Clostridium Difficile
Brief Title: Vancomycin for the Treatment of NAAT(+)/Toxin(-) C. Difficile
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Silvia Munoz-Price, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO00033844
Record Dates: First submitted 2019-01-21; First posted 2019-02-01 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium Difficile; Metabolomics; Vancomycin; Microbiome
MeSH Terms: conditions — Clostridium Infections | interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: Patients will be divided into 2 groups, one receiving oral vancomycin and the other placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: After enrollment, patients will be randomized to treatment with vancomycin 125 mg capsules by mouth every 6 hours for 14 days or to placebo with identical looking capsules for the same length of treatment. Block randomization will be used to assign patients to the treatment or placebo arms. Randomized assignments will be placed in sealed envelopes which will only be handled by the research pharmacist. Clinical providers, research team, and patients will remain blinded to allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug: Vancomycin Group (Active Comparator): Subjects will receive oral vancomycin capsules by mouth, 125 mg every 6 hours for 14 days.
  Interventions: Drug: Vancomycin Oral Capsule
- Drug: Placebo Group (Placebo Comparator): Subjects will receive a placebo oral capsule by mouth every 6 hours for 14 days. The placebo oral capsule is manufactured by Study Site's pharmacy to be identical in size, shape, color, appearance and taste as the drug comparator
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Vancomycin Oral Capsule — 125 mg capsules every 6 hours for 14 days.
  Other Names: Vancocin
  Arms: Drug: Vancomycin Group
Drug: Placebo Oral Capsule — Gelatin pill manufactured to mimic 125 mg Vancomycin oral capsule
  Arms: Drug: Placebo Group

SUMMARY:
This study proposes to:

1. Characterize the impact of oral vancomycin on C. difficile loads after end of treatment compared to a placebo group.
2. Determine the effect of oral vancomycin on structural and functional microbiome changes after end of treatment compared to a placebo group.
3. Characterize the impact of oral vancomycin against a placebo group on the daily frequency of loose stools by the end of treatment.

DETAILED DESCRIPTION:
Clostridium difficile infection (CDI) is considered the most frequent healthcare associated infection in the US, causing almost half a million cases per year with an estimated annual cost of 4.8 billion dollars. Despite the existence of a few treatment options against CDI, yearly attributable deaths are estimated at 29,300 in the US. From April 2014 to April 2016, Froedtert Health reported 899 CDIs. Over half of these events are NAAT (Nucleic Acid Amplification Test)(+)/EIA (Enzyme immunoassay)(-) events. To test for CDI, NAAT followed by EIA is used in a Multistep algorithmic testing in which a sensitive nucleic acid amplification test (NAAT) is followed by a specific toxin A and toxin B enzyme immunoassay (EIA) and are among the most accurate methods for Clostridium difficile infection (CDI) diagnosis. There is currently uncertainty on how to treat these CDI events.

The primary outcome of this randomized double blind controlled intervention trial will be changes in C. difficile (Clostridium difficile) loads between day 1 and day 14 and changes in C. difficile load between day 14 and day 28. Thirty patients with documented C. difficile will be randomized to either 14 days of vancomycin or placebo capsules. Block randomization will be used to assign patients to the treatment or placebo arms. Randomized assignments will be placed in sealed envelopes which will only be handled by the research pharmacist. Study related stool collections will be obtained on days 1, 7, 14, 21, and 28 (+/- 2days) [Day 1=first day study drug was administered]. Patients will be followed for 90 days starting on day 1. Patients unable to complete at least 7 days of study treatment will be removed from analysis and replaced.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age at time of consent.
* Presence of loose stools triggering clinical C. difficile NAAT/toxin EIA testing.
* Having both C. difficile NAAT (+) and C. difficile toxin EIA (-).
* Admitted outside the hematology-oncology unit.
* Must be willing to keep a study supplied drug diary

Exclusion Criteria:

* Presence of sepsis. Sepsis will be defined as a Sequential [Sepsis-related] Organ Failure Assessment (SOFA) score of 2 points or more as per 2016 definitions.
* Inability to take oral medications.
* Unwillingness or inability to provide written informed consent.
* Has a documented allergy to vancomycin.
* Has a documented life expectancy shorter than treatment course (14 days).
* Unwilling or unable to collect stool samples in the outpatient setting after discharge.
* Diagnosis of C. difficile colitis [NAAT(+) and toxin EIA(+)] in the preceding 3 months from enrollment.
* Received oral vancomycin during their current hospitalization, excluding empiric treatment given while pending C. difficile NAAT/toxin EIA results. Intravenous vancomycin is not an exclusion criterion.
* Women known to be pregnant or lactating during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Determine the change in C. difficile loads between the vancomycin vs. placebo group. | Day 1- Day 28
  Compare the impact of vancomycin vs placebo on changes in C. difficile load from stool samples collected on Day 1 to end-of-treatment (Day 14) and to Day 28 using quantitative Polymerase Chain Reaction (qPCR).
Determine the long-term persistence of C. difficile from the change in qPCR levels between the vancomycin vs. placebo group | Day 1 - Day 90
  Establish the long-term persistence of C. difficile by qPCR from stool samples collected at Day 1, 7, 14, 21, 28, and 90 between the vancomycin and placebo group.

SECONDARY OUTCOMES:
Characterize the change on structural alterations of the microbiome after end of treatment between the vancomycin vs. placebo groups through 16S rRNA sequencing. | Pre-treatment, Day 1 - Day 90 past the beginning of treatment
  Structural alterations of the microbiome after end of treatment will be determined using 16S rRNA sequencing from stool samples collected upon diagnosis, Days 1, 7, 14, 21, 28 & 90. Structural alterations will be defined according to the Shannon Diversity Index.
Measure the change in bile acids in the oral vancomycin vs. placebo groups by mass spectrometry. | Pre-treatment, Day 1 - Day 90 past the beginning of treatment
  Characterize the impact of oral vancomycin against placebo on functional microbiome changes after end of treatment by measuring bile acids. They will be measured via mass spectrometry using stool samples collected upon diagnosis, Days 1, 7, 14, 21, 28 & 90.
Measure the change in amino acids in the oral vancomycin vs. placebo groups by mass spectrometry. | Pre-treatment, Day 1 - Day 90 past the beginning of treatment
  Characterize the impact of oral vancomycin against placebo on functional microbiome changes after end of treatment by measuring amino acids. They will be measured via mass spectrometry using stool samples collected upon diagnosis, Days 1, 7, 14, 21, 28 & 90.
Measure the change in sugars in the oral vancomycin vs. placebo groups by mass spectrometry. | Pre-treatment, Day 1 - Day 90 past the beginning of treatment
  Characterize the impact of oral vancomycin against placebo on functional microbiome changes after end of treatment by measuring sugars. They will be measured via mass spectrometry using stool samples collected upon diagnosis, Days 1, 7, 14, 21, 28 & 90.
Measure the change in lipids from Day 1 to Day 90 in the oral vancomycin vs. placebo groups by mass spectrometry. | Pre-treatment, Day 1 - Day 90 past the beginning of treatment
  Characterize the impact of oral vancomycin against placebo on functional microbiome changes after end of treatment by measuring lipids. They will be measured via mass spectrometry using stool samples collected upon diagnosis, Days 1, 7, 14, 21, 28 & 90.
Measure the change in frequency of bowel movements in the oral vancomycin vs. placebo groups. | Day 1 - Day 90 past the beginning of treatment
  Characterize the impact of oral vancomycin against a placebo group on the daily frequency of bowel movements by the end of treatment. This scale goes from 0 to >20 in increments of 1. Data will be analyzed over time as a slope for each patient. The closer to 1 per 24 hours the better the outcome. Data will be obtained from patient self-reports using study questionnaires on Days 1, 7, 14, 21, 28 & 90.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Munoz-Price, M.D., Ph.D., Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Inc., Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Participant data to be shared would consist of age categories, genders, treatment groups, Clostridium difficile status, microbiome profile and metabolic profile. The data will be anonymized to prevent the identification of individual patients from the data provided. The data would be made available through contacting the principal investigator directly.